CLINICAL TRIAL: NCT00237302
Title: A Comparison of the Efficacy and Safety of Topiramate Versus Placebo for the Prophylaxis of Migraine in Pediatric Subjects
Brief Title: A Comparison of the Efficacy and Safety of Topiramate Versus Placebo in Preventing Migraine Headaches in Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ortho-McNeil Neurologics, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CR002662
Record Dates: First submitted 2005-10-07; First posted 2005-10-12 (Estimated); Last update posted 2011-05-19 (Estimated); Status verified 2010-04

CONDITIONS: Migraine
Keywords: pediatric migraine; migraine headache; migraine prophylaxis; migraine prevention; migraine
MeSH Terms: conditions — Migraine Disorders | interventions — Topiramate

INTERVENTIONS:
Drug: topiramate

SUMMARY:
The purpose of this study is to assess the safety and efficacy of topiramate as compared to placebo in preventing migraines in children.

DETAILED DESCRIPTION:
Pediatric migraine headache is a common cause of severe recurring headaches in children, especially children between the ages of 5 and 15 years. These headaches can be disabling and tend to interfere with a child's daily activities, such as going to school or playing with friends. Because pediatric migraine children tend to be misdiagnosed, they are often not treated effectively. Topiramate, an anti-seizure medication, has been shown to prevent migraines in adults, and it has been approved to treat seizures in children as young as 2 years of age as add-on treatment (used with another drug) and also can be used alone (monotherapy) in children as young as 10 years old. Since topiramate has already been studied in children, information about its safety in children is available. In this study, children with migraine headaches will be identified. It is not necessary for the child to have the migraine aura (having blurry vision; seeing flashing lights) to be included in this study. This is a randomized, double-blind, placebo-controlled study of Topiramate (or placebo) given for 4 to 5 months. An optional 3-month open-label extension (topiramate only; no placebo) will follow. The objective of the study is to demonstrate that topiramate is effective and safe when used to prevent migraine headaches (with or without aura) in children. Safety will be assessed throughout the study.

Topiramate sprinkle capsules (or placebo), starting at 15 milligrams per day for 1st week; increased to 30 milligrams per day for week 2; increased to 50 milligrams (in tablets) per day in week 3, then adjusted as needed to 2 to 3 milligrams/kilogram/day for the rest of study (140 days total).

ELIGIBILITY:
Inclusion Criteria:

* Children who have had several attacks of headaches that meet the International Headache Society Classification of pediatric migraine with or without aura (for example, headache lasts up to 48 hours, has a throbbing quality, is accompanied by nausea or sensitivity to light, is made worse by physical activity)
* Average of 3 to 10 migraine days per month for previous 3 months
* Weighs more than 20 kilograms (44 pounds)
* Able to swallow a tablet whole (without crushing it)

Exclusion Criteria:

* Took topiramate previously to prevent migraines but it was not effective
* Had to stop taking topiramate because of side effects
* Presence of cluster headaches, migraine aura without headache
* Had taken any medications for migraine prevention within 2 weeks before study start
* Presence of active liver disease or abnormal kidney function

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 162 (Actual)
Dates: Start 2001-07; Study Completion 2003-09 (Actual)

PRIMARY OUTCOMES:
Number of migraine days per month (28 days) during the double-blind treatment period relative to the prospective baseline period.

SECONDARY OUTCOMES:
Monthly rates of migraine episodes, non-migraine headache episodes, and total headache days; percentage of treatment responders; severity and duration of migraines; frequency and severity of associated migraine symptoms, and use of rescue medicines.

CONTACTS AND LOCATIONS:
Overall Officials: Ortho McNeil Neurologics, Inc. Clinical Trial, Study Director — Ortho-McNeil Neurologics, Inc.

REFERENCES:
- See also: A Comparison of the Efficacy and Safety of Topiramate Versus Placebo for the Prophylaxis of Migraine in Pediatric Subjects — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=916&filename=CR002662_CSR.pdf